CLINICAL TRIAL: NCT07338162
Title: Is Serial Casting a Valid Option for Management of Lower Limb Deformities in Patient With Spastic Cerebral Palsy (Equinus - Equinovarus)?
Brief Title: Is Serial Casting a Valid Option for Management of Lower Limb Deformities in Patient With Spastic Cerebral Palsy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdou Mohamed Dawood, Orthopaedic Surgery specialist at Al-Helal Hospital, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-97-2023
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Serial Casting; Management; Lower Limb Deformities; Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Children with spastic cerebral palsy who is subjected to a selected physical therapy program once a day/3 times a week for three successive weeks mainly consisted of stretching and strengthening exercises, weight bearing, balance, proprioception, and ambulation training.
  Interventions: Other: Physical therapy program
- Group B (Experimental): Children with spastic cerebral palsy who is additionally subjected to three consecutive casts applied for five days each and will be removed in the last two days in each week to conduct the same selected physical therapy program.
  Interventions: Other: Three consecutive casts + Physical therapy program

INTERVENTIONS:
Other: Physical therapy program — Children with spastic cerebral palsy who is subjected to a selected physical therapy program once a day/3 times a week for three successive weeks mainly consisted of stretching and strengthening exercises, weight bearing, balance, proprioception, and ambulation training.
  Arms: Group A
Other: Three consecutive casts + Physical therapy program — Children with spastic cerebral palsy who is additionally subjected to three consecutive casts applied for five days each and will be removed in the last two days in each week to conduct the same selected physical therapy program.
  Arms: Group B

SUMMARY:
This study aimed to evaluate the effectiveness of serial casting as a modality of management of lower limb deformities in patients with spastic cerebral palsy (equinous - equinovarus).

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is classified as a group of postural and motor disorders caused by a non-progressive lesion to the developing brain, acquired before the age of two. Among the different types of CP, spastic CP is the most common form consisting of approximately 85.8% of diagnoses.

Current clinical management of spasticity and contracture in the lower limb includes conservative approaches such as the use of physiotherapy, orthoses, casting and splinting. Other commonly used invasive strategies for spasticity and contracture management include neurotoxin injections such as botulinum toxin A (BTX-A) and intrathecal baclofen, as well as surgery such as selective dorsal rhizotomy (SDR) and various corrective orthopaedic operations including tendon lengthening procedures and single-event multilevel surgeries (SEMLS).

ELIGIBILITY:
Inclusion Criteria:

* Patients from 3 to 12 years old.
* Both sex.
* Spastic cerebral palsy patients with true equinous.
* Modified Ashworth Scale score of 2 or 3 in the plantar flexor muscle complex.
* Gross Motor Functional Classification System Level I, II & III.

Exclusion Criteria:

* Patients with bony joint limitation.
* Previous surgeries (tendon lengthening).
* Patients received Botulinum toxin A injections in the last six months.
* Patients with apparent equinus as a compensation for knee or hip flexion while dorsiflexion range is preserved at the lower extremity.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of ankle range of motion | 3 months after the procedure
  Ankle range of motion was assessed.

SECONDARY OUTCOMES:
Tone of the calf muscle | 3 months after the procedure
  Tone of the calf muscle was measured.
Detection of ankle kinematics during gait | 3 months after the procedure
  The children will be instructed to walk and videos were taken from the side, only five sections were tested to evaluate ankle kinematics and knee position in relation to ankle (initial foot contact, foot contact at mid stance, timing of heel rise, knee position in mid stance, degree of change) with a total score of 14 on each limb.
Incidence of true equinous in patients with spastic cerebral palsy | 3 months after the procedure
  Incidence of true equinous in patients with spastic cerebral palsy was assessed.
Modified Ashworth Scale (MAS) score | 3 months after the procedure
  The Modified Ashworth Scale (MAS) score is a widely used measurement tool, and it is scored as follows: 0, no increase in muscle tone; 1, slight increase in muscle tone at the end of the range of motion; 2, slight increase in muscle tone through less than half of the range of motion; 3, more marked increase in muscle tone through most of the range of motion; 4, considerable increase in muscle tone; and 5, joint is rigid.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.